CLINICAL TRIAL: NCT02233946
Title: Computerized Alcohol Screening for Children and Adolescents (cASCA) in Primary Care
Acronym: cASCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Principal Investigator, Sion Kim Harris, Co-Director, Center for Adolescent Substance Abuse Research, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P00004862; 1R01AA021904-01 (NIH)
Record Dates: First submitted 2014-08-19; First posted 2014-09-09 (Estimated); Results first posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-02

CONDITIONS: Prevention Harmful Effects
Keywords: Substance Abuse; Prevention; Youth; Alcohol; Drugs
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- screening w/ computer brief intervention (Experimental): screening with computer-facilitated brief intervention
  Interventions: Behavioral: computer-facilitated brief intervention
- Screening with Treatment as Usual (No Intervention): Screening with Treatment as Usual

INTERVENTIONS:
Behavioral: computer-facilitated brief intervention — Immediate feedback to patient of screening results and risk for substance use problem, followed by 11 pages of science and true-life stories about health risks of adolescent substance use. Screening results then go to provider who reviews them with patient and gives brief counseling, and refers to an online motivational enhancement therapy intervention for patients at moderate/high risk for substance use problems.
  Arms: screening w/ computer brief intervention

SUMMARY:
The purpose of this study is to assess the psychometric properties of a brief screening questionnaire for alcohol problems among 9- to 18-year-old patients in pediatricians' offices, and to pilot test a personalized, computer-facilitated brief intervention delivered on a tablet computer and by the provider based on screening results.

DETAILED DESCRIPTION:
The primary goal of this project is to develop a computerized screening program for primary care offices that is based on the NIAAA's new Alcohol Screening Guide for Children and Adolescents and assess its psychometric properties among nine- to 18-yr-old primary care patients. There is substantial evidence supporting the effectiveness of screening and brief intervention among adult primary care patients, primarily in the reduction of harmful drinking. However, there have been few studies of alcohol screening and brief intervention conducted among adolescents seen in busy primary care settings. This project will develop and validate a new computerized Alcohol Screening for Children and Adolescents (cASCA) program which incorporates the age-specific screening questions of the NIAAA Guide and includes the CRAFFT and AUDIT as secondary risk/problem assessments. We will add tobacco screening because tobacco use is the leading cause of cancer-related mortality in the US as well as screening for marijuana and other drug use so as to create a comprehensive screening instrument that includes all major substances that adolescents use.

Additionally, the NIAAA guide recommends that providers deliver a brief intervention in response to the screening results. Therefore, a secondary aim of this project will be to pilot-test a computer-facilitated Brief Intervention component using a randomized design comparing three groups: 1) screening with treatment as usual [cASCA/TAU]; 2) screening with the computer-facilitated brief intervention [cASCA/BI]. The BI component consists of patients viewing on the computer, immediately after the screening, their score and level of risk for a substance use problem, as well as several interactive pages of science and true-life stories about the health risks of substance use. Clinicians are then given the screen results and suggested talking points for a few minutes of brief counseling during the visit.

Hypothesis: Among 9- to 18-year-old primary care patients, those receiving cASCA/BI will have lower rates of any alcohol use, days of alcohol use, drinks per drinking day, and days of heavy episodic drinking, at 3, 6, 9 and 12-months follow-up than those receiving treatment as usual.

ELIGIBILITY:
Inclusion Criteria:

* access to computer and email address
* available and willing to complete all follow ups by email or phone
* medically and emotionally stable
* can read and understand English

Exclusion Criteria:

* Patient has already participated in this study

Ages: 9 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 871 (Actual)
Dates: Start 2015-01; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John R Knight, MD, Principal Investigator — Boston Children's Hospital; Sion K Harris, PhD, Principal Investigator — Boston Children's Hospital
Locations (5):
- United States (5):
  - Tufts Medical Center, Boston, Massachusetts
  - Boston Childrens Primary Care Center, Boston, Massachusetts
  - Longwood Pediatrics, Boston, Massachusetts
  - East Boston Neighborhood Health Center, East Boston, Massachusetts
  - Lexington Pediatrics, Lexington, Massachusetts

REFERENCES:
- [Background] Harris SK, Csemy L, Sherritt L, Starostova O, Van Hook S, Johnson J, Boulter S, Brooks T, Carey P, Kossack R, Kulig JW, Van Vranken N, Knight JR. Computer-facilitated substance use screening and brief advice for teens in primary care: an international trial. Pediatrics. 2012 Jun;129(6):1072-82. doi: 10.1542/peds.2011-1624. Epub 2012 May 7. PMID 22566420
- See also: Center for Adolescent Substance Abuse Research — http://www.ceasar.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Computerized Screening w/ Provider Brief Intervention (cSBI): cSBI consists of adolescents self-administering on a tablet computer a screening questionnaire prior to seeing their provider. The computer program then immediately provides adolescents with personalized feedback, followed by brief psychoeducation illustrating the health-related risks of substance use. Providers then login to the tablet computer to access a Clinician Report Form which presents the patient's screening results, as well as discussion prompts to guide a few minutes of Motivational Interviewing-based brief counseling during the visit.
- Computerized Screening With Treatment as Usual (TAU): The comparison group also completed the computerized screening tool. However, this group did not receive any feedback or psychoeducation, and their providers did not receive the screening results. During the visit, adolescents in this group received treatment as usual.
Period: Baseline
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Started | 628 (Allocated to and received the intervention) | 243 (Allocated to and received usual care)
Completed | 626 (Completed baseline assessment) | 243 (Completed baseline assessment)
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0
Period: Immediate Post-visit Questionnaire
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Started | 626 | 243
Completed | 624 | 243
Not Completed | 2 | 0
Period: 3-months Follow-up
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Started | 624 | 243
Completed | 571 | 214
Not Completed | 53 | 29
Not completed — Lost to Follow-up | 53 | 29
Period: 6-months Follow-up
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Started | 571 | 214
Completed | 550 | 212
Not Completed | 21 | 2
Not completed — Lost to Follow-up | 21 | 2
Period: 9-month Follow-up
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Started | 550 | 212
Completed | 530 | 201
Not Completed | 20 | 11
Not completed — Lost to Follow-up | 20 | 11
Period: 12-month Follow-up
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Started | 530 | 201
Completed | 502 | 190
Not Completed | 28 | 11
Not completed — Lost to Follow-up | 28 | 11

BASELINE CHARACTERISTICS:
Population: 12- to 18-year-olds arriving for their annual well-visit at participating pediatric practices
Groups:
- Total: Total of all reporting groups
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 626 | 243 | 869
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  years
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline | 16.3 (1.3) | 16.5 (1.3) | 16.4 (1.3)
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline | 14.1 (1.8) | 14.5 (1.7) | 14.3 (1.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Female | 80 | 34 | 114
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Male | 68 | 29 | 97
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Female | 236 | 91 | 327
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Male | 242 | 89 | 331
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Non-Hispanic White | 69 | 36 | 105
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Hispanic | 40 | 15 | 55
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Other or multirace | 39 | 12 | 51
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Non-Hispanic White | 203 | 79 | 282
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Hispanic | 143 | 58 | 201
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Other or multirace | 132 | 43 | 175
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 626 | 243 | 869
In grades 9-12 [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 141 | 60 | 201
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 7 | 3 | 10
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 197 | 100 | 297
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 281 | 80 | 361
Lives with two parents in home [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 103 | 41 | 144
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 45 | 22 | 67
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 380 | 143 | 523
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 98 | 37 | 135
Parent highest education level is college graduate or higher [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 100 | 44 | 144
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 48 | 19 | 67
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 306 | 108 | 414
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 172 | 72 | 244
Saw a pediatrician at visit [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 128 | 50 | 178
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 20 | 13 | 33
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 412 | 152 | 564
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 66 | 28 | 94
Saw a female practitioner [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 99 | 50 | 149
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 49 | 13 | 62
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 321 | 117 | 438
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 157 | 63 | 220
Had 6 or more prior visits with practitioner [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 90 | 33 | 123
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 58 | 30 | 88
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 284 | 106 | 390
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 194 | 74 | 268
Had CRAFFT score of 2 or greater [Count of Participants; unit: Participants] — Score of >=2 suggests a serious problem and warrants clinical attention. C-Have you ever ridden in a CAR driven by someone (including yourself) who was "high" or had been using alcohol or drugs? R-Do you ever use alcohol or drugs to RELAX, feel better about yourself, or fit in? A-Do you ever use alcohol or drugs while you are by yourself, or ALONE? F-Do you ever FORGET things you did while using alcohol or drugs? F-Do your family or FRIENDS ever tell you that you should cut down on your drinking or drug use? T-Have you ever gotten into TROUBLE while you were using alcohol or drugs? Population: Participants who reported past-12-month use of alcohol or other drugs at baseline
  Participants
    Yes: number analyzed (Participants) | 148 | 63 | 211
    Yes | 41 | 18 | 59
    No: number analyzed (Participants) | 148 | 63 | 211
    No | 107 | 45 | 152
Hung out with friends who use alcohol/drugs [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 131 | 57 | 188
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 17 | 6 | 23
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 169 | 82 | 251
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 309 | 98 | 407
Has substance-involved siblings [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 59 | 23 | 82
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 89 | 40 | 129
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 40 | 10 | 50
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 438 | 170 | 608
Has substance-involved parents/guardians [Count of Participants; unit: Participants] — Population: We conducted analyses stratified by past-12-month use of any alcohol or other drugs reported at baseline
  Participants
    Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 148 | 63 | 211
    Participants who reported past-12-month use of alcohol or other drugs at baseline: Yes | 25 | 10 | 35
    Participants who reported past-12-month use of alcohol or other drugs at baseline: No | 123 | 53 | 176
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 478 | 180 | 658
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: Yes | 27 | 8 | 35
    Participants who reported no past-12-month use of alcohol or other drugs at baseline: No | 451 | 172 | 623

OUTCOME MEASURES:

1. Primary Outcome: Time to First Post-visit Drinking Day
Description: Median (and interquartile range) for times to first use for the cSBI and Treatment As Usual (TAU) groups
Time Frame: 12-months follow-up
Population: Stratified: Participants who reported past-12-month use of alcohol or other drugs at baseline vs. Participants who reported no past-12-month use of alcohol or other drugs at baseline
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Number analyzed (Participants) | 570 | 212
days
  Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 114 | 46
  Participants who reported past-12-month use of alcohol or other drugs at baseline | 97 [51 to 222] | 44 [21 to 143]
  Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 456 | 166
  Participants who reported no past-12-month use of alcohol or other drugs at baseline | 366 [338 to 366] | 366 [334 to 366]
Statistical Analysis 1: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants who reported past-12-month use of alcohol or other drugs at baseline; Test type: Superiority; Cox Proportional Hazard = 0.69, 95% CI 2-sided [0.47 to 1.02]
Statistical Analysis 2: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants who reported no past-12-month use of alcohol or other drugs at baseline; Test type: Superiority; Cox Proportional Hazard = 0.87, 95% CI 2-sided [0.57 to 1.31]

2. Primary Outcome: Time to First Post-visit Heavy Episodic Drinking Day
Description: The number of days post-visit to first reported heavy episodic drinking day
Time Frame: 12-months follow-up
Population: Participants who reported past-12-month use of alcohol or other drugs at baseline
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Number analyzed (Participants) | 114 | 46
days | 366 [124 to 366] | 213 [51 to 366]
Statistical Analysis 1: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants who reported past-12-month use of alcohol or other drugs at baseline; Test type: Superiority; Cox Proportional Hazard = 0.66, 95% CI 2-sided [0.40 to 1.10]

3. Secondary Outcome: Time to First Post-visit Cannabis Use Day
Description: The number of days post-visit to first reported cannabis use day.
Time Frame: 12-months follow-up
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Number analyzed (Participants) | 516 | 191
Days
  Participants who reported past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 60 | 25
  Participants who reported past-12-month use of alcohol or other drugs at baseline | 101 [33 to 226] | 83 [27 to 152]
  Participants who reported no past-12-month use of alcohol or other drugs at baseline: number analyzed (Participants) | 456 | 166
  Participants who reported no past-12-month use of alcohol or other drugs at baseline | 366 [366 to 366] | 366 [366 to 366]
Statistical Analysis 1: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Test type: Superiority — Participants who reported past-12-month use of alcohol or other drugs at baseline; Cox Proportional Hazard = 0.62, 95% CI 2-sided [0.41 to 0.94]
Statistical Analysis 2: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants who reported no past-12-month use of alcohol or other drugs at baseline; Test type: Superiority; Cox Proportional Hazard = 0.76, 95% CI 2-sided [0.44 to 1.32]

4. Secondary Outcome: Past-3-month Riding Risk
Description: Self-reported riding in the past 3 months with a driver who had been drinking or using other drugs, stratified by reported riding risk in the past 3 months at baseline
Time Frame: 12 months follow-up
Population: Participants with riding risk at baseline vs. those with no riding risk at baseline. (Differences in number of participants analyzed at each follow-up time point is due to number of survey respondents at that time point. For example, in the cSBI group at baseline, 64 participants reported having riding risk. At 3 months follow-up, 44 of those completed a survey, and 20 of those 44 reported having riding risk at the 3-months follow-up.)
Measure: Number; unit: participants
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
Number analyzed (Participants) | 625 | 243
participants
  Riding risk at baseline : Baseline, No.: number analyzed (Participants) | 64 | 35
  Riding risk at baseline : Baseline, No. | 64 | 35
  Riding risk at baseline : 6 months: number analyzed (Participants) | 44 | 21
  Riding risk at baseline : 6 months | 20 | 12
  Riding risk at baseline : 9 months: number analyzed (Participants) | 39 | 21
  Riding risk at baseline : 9 months | 16 | 13
  Riding risk at baseline : 12 months: number analyzed (Participants) | 45 | 19
  Riding risk at baseline : 12 months | 18 | 13
  No riding risk at baseline : Baseline, No.: number analyzed (Participants) | 561 | 208
  No riding risk at baseline : Baseline, No. | 561 | 208
  No riding risk at baseline : 6 months: number analyzed (Participants) | 429 | 158
  No riding risk at baseline : 6 months | 35 | 19
  No riding risk at baseline : 9 months: number analyzed (Participants) | 419 | 163
  No riding risk at baseline : 9 months | 33 | 10
  No riding risk at baseline : 12 months: number analyzed (Participants) | 452 | 168
  No riding risk at baseline : 12 months | 28 | 11
Statistical Analysis 1: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants with riding risk at baseline: Adjusted Relative Risk Ratio (ARRR) of past-3-month riding risk at 6 months follow-up, cSBI vs. TAU; Test type: Superiority; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.50 to 1.34]
Statistical Analysis 2: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants with riding risk at baseline: Adjusted Relative Risk Ratio (ARRR) of past-3-month riding risk at 9 months follow-up, cSBI vs. TAU; Test type: Superiority; Risk Ratio (RR) = 0.73, 95% CI 2-sided [0.44 to 1.19]
Statistical Analysis 3: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants with riding risk at baseline: Adjusted Relative Risk Ratio (ARRR) of past-3-month riding risk at 12 months follow-up, cSBI vs. TAU; Test type: Superiority; Risk Ratio (RR) = 0.58, 95% CI 2-sided [0.37 to 0.91]
Statistical Analysis 4: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants with no riding risk at baseline: Adjusted Relative Risk Ratio (ARRR) of past-3-month riding risk at 6 months follow-up, cSBI vs. TAU; Test type: Superiority; Risk Ratio (RR) = 0.72, 95% CI 2-sided [0.43 to 1.23]
Statistical Analysis 5: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants with no riding risk at baseline: Adjusted Relative Risk Ratio (ARRR) of past-3-month riding risk at 9 months follow-up, cSBI vs. TAU; Test type: Superiority; Risk Ratio (RR) = 1.33, 95% CI 2-sided [0.67 to 2.66]
Statistical Analysis 6: Comparison: Computerized Screening w/ Provider Brief Intervention (cSBI) vs Computerized Screening With Treatment as Usual (TAU); Participants with no riding risk at baseline: Adjusted Relative Risk Ratio (ARRR) of past-3-month riding risk at 12 months follow-up, cSBI vs. TAU; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.50 to 1.99]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Computerized Screening w/ Provider Brief Intervention (cSBI) | Computerized Screening With Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 0/626 | 0/243
Serious Adverse Events (participants affected / at risk) | 0/626 | 0/243
Other Adverse Events (participants affected / at risk) | 0/626 | 0/243

LIMITATIONS AND CAVEATS:
Same practitioners delivering both the CSBI and UC may have contaminated UC arm; only group difference we could assure was the CRAFFT screen. Relied on patients' reporting of intervention; did not obtain independent observations of practitioner behaviors. Relied on self-report. Unable to examine effects on use of certain drugs (low prevalence). Did not collect parents' views of CSBI system.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-11-13): https://cdn.clinicaltrials.gov/large-docs/46/NCT02233946/Prot_SAP_000.pdf